CLINICAL TRIAL: NCT07002528
Title: The Effectiveness of Sweet Solution Versus Cryotherapy in Reducing Pain During Administration of Local Anesthesia Among Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Manwa Ayed, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ِA0203024PP
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pain
Keywords: Dental pain; Anesthesia; Sucrose; Cryotherapy; Topical anesthesia
MeSH Terms: conditions — Pain; Toothache | interventions — sodium lactobionate sucrose solution; Cryotherapy; Anesthesia

STUDY DESIGN:
Intervention Model Description: Selected children will be divided randomly into 3 groups:
  Sucrose group (Group I). Cryotherapy group (Group II). Control group topical anesthesia (Group III).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- apply treatment with sucrose solution as analgesic before admenistration of local anesthesia (Experimental)
  Interventions: Behavioral: sucrose solution
- apply treatment with cryotherapy as analgesic before admenistration of local anesthesia (Experimental)
  Interventions: Behavioral: Cryotherapy
- apply normal treatment with topical anesthesia before admenistration of local anesthesia (Experimental)
  Interventions: Behavioral: topical anesthesia

INTERVENTIONS:
Behavioral: sucrose solution — apply sucrose solution to evaluate pain among local anesthesia
  Arms: apply treatment with sucrose solution as analgesic before admenistration of local anesthesia
Behavioral: Cryotherapy — apply cryotheraby to evaluate pain among local anesthesia
  Arms: apply treatment with cryotherapy as analgesic before admenistration of local anesthesia
Behavioral: topical anesthesia — apply topical anesthesia to evaluate pain among local anesthesia
  Arms: apply normal treatment with topical anesthesia before admenistration of local anesthesia

SUMMARY:
the porpose of study to assess The Effectiveness of Sweet Solution Versus Cryotherapy in Reducing Pain During Administration of Local Anesthesia Among Children

DETAILED DESCRIPTION:
This study to assess The Effectiveness of Sweet Solution Versus Cryotherapy in Reducing Pain During Administration of Local Anesthesia Among Children

ELIGIBILITY:
Inclusion Criteria:

1. Children with behavior rating score 2,3 or 4 of Frankl's behavior rating scale
2. children aged 6-11 years requiring dental injections for pulpectomy, root canal treatment, or extraction procedures for primary and permanent mandibular molars.

Exclusion criteria:

1. Allergy to lidocaine
2. Redness at the site of injection؛ and a history of abscess, sinus tract, or fistula associated with the teeth.
3. Children with special health care needs.
4. Children suffering from systemic diseases.
5. Extremely uncooperative children.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
VAS | up to twelve weeks
  a simple, 10-cm line used to measure pain intensity in children, with word anchors at each end like "no pain" and "worst possible pain". Children are asked to mark the point on the line that represents their pain level, and the distance from the "no pain" anchor is used to calculate the score. While VAS is generally considered reliable for children 5 years and older, some studies suggest younger children may struggle with the conceptual complexity.
FLACC scale | up to twelve weeks
  a behavioral pain assessment tool used for children, especially those who cannot verbally express their pain. It stands for Face, Legs, Activity, Cry, and Consolability. The FLACC scale is used to assess pain in infants and children from birth and older, including those with developmental delays. It's a way to understand pain by observing facial expressions and behavioral patterns. Each of the five categories is scored on a 0-2 scale, resulting in a total pain score from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Manwa Ahmed Ayed, Master, Study Chair — Researcher of Pediatric Dentistry Faculty of Dentistry Mansoura University; Salwa M Awad, prof, Study Director — Prof. of Pediatric Dentistry and Dental Public Health Faculty of Dentistry Mansoura University; Ahmed Hamdy Wahba, Assistant professor, Study Director — assistant Prof. of Pediatric Dentistry and Dental Public Health Faculty of Dentistry Mansoura University
Locations (1):
- Mansoura university, Al Mansurah, Dakahilia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study protocol to other researcher
Supporting Information: Study Protocol
Time Frame: within 6 month
Access Criteria: for any one